CLINICAL TRIAL: NCT07224178
Title: Left Atrial Strain: A Biomarker for Cryptogenic Stroke Prevention
Brief Title: Left Atrial Strain and Cryptogenic Stroke
Acronym: LAS-ESUS
Status: Recruiting | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Leyla Sade, Professor of Medicine, University of Pittsburgh
Other Study IDs: STUDY25010088
Record Dates: First submitted 2025-10-28; First posted 2025-11-04 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Ischemic Stroke, Cryptogenic; Ischemic Stroke, Embolic; Hemorrhagic Stroke; Embolic Stroke of Undetermined Source; Recurrent Ischemic Stroke
Keywords: stroke; embolic stroke of undetermined source; speckle-tracking echocardiography; left atrial cardiomyopathy; left atrial strain; recurrent ischemic stroke; new-onset atrial fibrillation
MeSH Terms: conditions — Ischemic Stroke; Hemorrhagic Stroke; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cryptogenic Stroke Cohort: Subjects in sinus rhythm who had a diagnosis of ischemic embolic stroke in whom no clear embolic source was identified after standard diagnostic evaluation (TOAST classification: Embolic Stroke of Undetermined Source) and who had transthoracic echocardiography (TTE) as part of the stroke work up will constitute the first group.
- Non-Cryptogenic Stroke Cohort (Comparator Group): Subjects in sinus rhythm who had a non-cryptogenic stroke (e.g., large artery atherosclerosis, small vessel disease, hemorrhagic) and who underwent transthoracic echocardiography as part of the clinical stroke workup.
  This group will serve as a comparator for the primary analysis to determine whether LA strain determines cryptogenic stroke among other stroke subtypes.

SUMMARY:
Cryptogenic stroke is a type of stroke in which the cause of the blood clot cannot be identified, leaving many patients without a clear treatment plan and at high risk for another stroke. Current medical guidelines recommend blood-thinning medication (anticoagulation) only when atrial fibrillation (AF) -an irregular heart rhythm- can be documented. However, AF may occur silently and remain undetected. Long term implantable (placed invasively under the skin) devices may be needed to capture these episodes.

AF is known to develop from disease of the left atrium, the upper chamber of the heart that receives blood from the lungs. When the left atrium does not contract normally, blood flow may slow down, increasing the risk of clot formation. Nowadays, the left atrial (LA) function can be quantified precisely using a noninvasive ultrasound technique called strain imaging.

This study aims to determine whether reduced LA function is associated with cryptogenic stroke and its recurrence even when AF is not observed. If such an association is confirmed, LA strain could serve as a new biomarker to identify patients at risk, earlier than the development of overt AF, enhance preventive measures to reduce recurrent strokes. Because echocardiographic strain imaging is safe, cost-effective, and widely available, it may become an important tool for improving care in this high-risk population.

DETAILED DESCRIPTION:
Cryptogenic stroke accounts for nearly one-third of ischemic strokes, yet its underlying mechanism often remains unidentified, leaving patients without targeted therapy. Atrial fibrillation (AF) is detected up to one third of cryptogenic strokes, but its detection frequently requires prolonged monitoring due to subclinical paroxysmal episodes. Increasing evidence suggests that structural and functional abnormalities of the left atrium (LA) precede AF and contribute to thromboembolic risk independently of rhythm disturbances.

This multicenter retrospective study aims to determine whether impaired LA strain, a sensitive echocardiographic measure of atrial function, is associated with cryptogenic stroke and can predict recurrent events. Echocardiographic images of the patients who were referred to the echocardiography laboratory as part of stroke work up will be analyzed offline, using standardized speckle-tracking software. De-identified clinical and imaging data will be collected in the central core laboratory at the University of Pittsburgh for uniform analysis and validation.

By establishing LA strain as a biomarker of atrial cardiopathy and cryptogenic stroke risk, this study seeks to bridge the current gap between stroke classification and management. Demonstrating the independent association between LA dysfunction and cryptogenic stroke and the recurrence of cryptogenic stroke independently of AF could support the use of LA strain as a risk marker to for monitoring patient and developing preventive strategies such as anticoagulation without documented AF. Hence, our findings may improve preventive care and reduce the burden of disabilities due to cryptogenic stroke.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age > 18 years and < 80 years) who had a complete transthoracic echocardiography (TTE) exam at the University of Pittsburgh Medical Center (UPMC) Presbyterian Echocardiography Lab with a referral diagnosis of suspected stroke.

  2- Patients with an established diagnosis of stroke by stroke neurologists.

  3- Patients in sinus rhythm documented at the time of referral.

  4- Availability of adequate echocardiographic images for strain quantification.

  5- Clinical follow-up data available for evaluation of study endpoints, including stroke recurrence, atrial fibrillation development, and mortality.

  6- Patients from collaborating centers will be included with de-identified echocardiographic images and clinical data meeting the above criteria.

Exclusion Criteria:

Incomplete or technically difficult transthoracic echocardiography (TTE) studies and studies from subjects younger than 18 years of age will be excluded. Additional exclusion criteria include:

1- Pre-existing atrial fibrillation (AF): Patients with a documented history AF prior to the index echocardiography study will be excluded because it is well established that AF justifies cryptogenic stroke requiring anticoagulation.

2 -Structural heart disease: Patients with significant structural abnormalities, such as moderate or severe mitral stenosis, moderate or severe mitral regurgitation, prosthetic heart valves, devices in the left atrium, atrial septal defect or patent foramen ovale will be excluded as these conditions are known causes of stroke and abnormal left atrial function.

3- Coagulopathy: Patient having disease leading to hypercoagulable (thrombus formation) state will be excluded (presence of cancer, antiphospholipid antibodies, hematological diseases).

4- Inadequate clinical follow-up: Patients with insufficient follow-up data or missing medical records that preclude evaluation of study endpoints (e.g., stroke recurrence, AF development) will be excluded unless death is documented.

5- Poor image quality for strain analysis: Patients having echo exams with inadequate image quality that prevent reliable strain quantification will be excluded.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be selected from adult patients evaluated for stroke at the University of Pittsburgh Medical Center (UPMC) and collaborating university hospitals that serve as tertiary care centers with established cardiovascular imaging programs.
  Only subjects who have already undergone transthoracic echocardiography as part of their stroke workup, and who have clinical and imaging data available for retrospective analysis will be included.
  The UPMC will provide both the data collection platform -REDCap- and Echocardiography Core Laboratory for centralized image analysis.
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2025-12-17 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Correlation between left atrial strain (percent deformation) and the rate of cryptogenic stroke | Baseline
  Quantitative left atrial (LA) strain (% deformation), measured by speckle-tracking echocardiography from transthoracic echocardiograms obtained during stroke workup, will be compared with the rate of cryptogenic stroke.

SECONDARY OUTCOMES:
Prediction of recurrent cryptogenic stroke by left atrial strain (percent deformation) | Up to 1 year from date of index transthoracic echocardiography.
  The number of recurrent cryptogenic stroke events during follow-up, as assessed by left atrial (LA) strain (% deformation) quantified at baseline echocardiogram.
Incidence of cardiovascular and cerebrovascular mortality among patients with impaired LA strain (percent deformation) | Up to 1 year from date of index transthoracic echocardiography.
  The number of cardiovascular and cerebrovascular mortality during follow-up, as assessed by left atrial (LA) strain (% deformation) quantified at baseline echocardiogram.
Incidence of newly detected atrial fibrillation among patients with impaired LA strain | Up to 1 year from date of index transthoracic echocardiography.
  The number of new-onset atrial fibrillation during follow-up, as assessed by left atrial (LA) strain (% deformation) quantified at baseline echocardiogram.

CONTACTS AND LOCATIONS:
Overall Officials: Leyla E Sade, MD, Principal Investigator — University of Pittsburgh Medical Center
Locations (1):
- UPMC Presbyterian, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) collected in this study, including baseline characteristics, clinical outcomes, and left atrial strain measurements, will be shared. Data will be available upon reasonable request for researchers conducting methodologically sound studies that align with the objectives of this research.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: IPD and supporting documents will be available starting 6 months after publication of the primary results and will remain accessible for 5 years thereafter.
Access Criteria: Access to the dataset will be granted to researchers upon submission of a formal request, outlining the study objectives and analysis plan. Approval will be contingent upon compliance with ethical guidelines, data privacy regulations, and institutional review board (IRB) requirements. Researchers will be required to sign a data-sharing agreement (DSA) before receiving access with the University of Pittsburgh..

REFERENCES:
- [Background] Maheshwari A, Norby FL, Inciardi RM, Wang W, Zhang MJ, Soliman EZ, Alonso A, Johansen MC, Gottesman RF, Solomon SD, Shah AM, Chen LY. Left Atrial Mechanical Dysfunction and the Risk for Ischemic Stroke in People Without Prevalent Atrial Fibrillation or Stroke : A Prospective Cohort Study. Ann Intern Med. 2023 Jan;176(1):39-48. doi: 10.7326/M22-1638. Epub 2022 Dec 20. PMID 36534978
- [Background] Masini G, Wang W, Ji Y, Eaton A, Inciardi RM, Soliman EZ, Passman RS, Solomon SD, Shah AM, De Caterina R, Chen LY. Markers of Left Atrial Myopathy: Prognostic Usefulness for Ischemic Stroke and Dementia in People in Sinus Rhythm. Stroke. 2025 Apr;56(4):858-867. doi: 10.1161/STROKEAHA.124.047747. Epub 2025 Mar 7. PMID 40052267
- [Background] Sade LE, Keskin S, Can U, Colak A, Yuce D, Ciftci O, Ozin B, Muderrisoglu H. Left atrial mechanics for secondary prevention from embolic stroke of undetermined source. Eur Heart J Cardiovasc Imaging. 2022 Feb 22;23(3):381-391. doi: 10.1093/ehjci/jeaa311. PMID 33206942
- [Background] Sade LE, Faletra FF, Pontone G, Gerber BLM, Muraru D, Edvardsen T, Cosyns B, Popescu BA, Klein A, Marwick TH, Cameli M, Saric M, Thomas L, Ajmone Marsan N, Fontes-Carvalho R, Podlesnikar T, Fontana M, La Gerche A, Petersen SE, Moharem-Elgamal S, Bittencourt MS, Vannan MA, Glikson M, Peichl P, Cochet H, Stankovic I, Donal E, Thomas D, Marta RS. The role of multi-modality imaging for the assessment of left atrium and left atrial appendage: a clinical consensus statement of the European Association of Cardiovascular Imaging (EACVI), European Heart Rhythm Association (EHRA) of the European Society of Cardiology (ESC). Eur Heart J Cardiovasc Imaging. 2025 Mar 3;26(3):385-413. doi: 10.1093/ehjci/jeaf014. PMID 39812172
- [Background] Clark A, Ferkh A, Vandenberg J, Elhindi J, Thomas L. Altered left atrial metrics in patients with cryptogenic stroke: A systematic review and meta-analysis. Eur J Clin Invest. 2024 Jun;54(6):e14175. doi: 10.1111/eci.14175. Epub 2024 Feb 2. PMID 38308431
- [Background] Ozbay B, Rearick C, Satyavolu BS, Soman P, Wong TC, Starr M, Pillai B, Zhu J, Azhar AZ, Katz WE, Sade LE. Primary Left Atrial Cardiopathy in Transthyretin Amyloidosis Cardiomyopathy by Multimodality Imaging: Implications for Thrombotic Events. JACC Cardiovasc Imaging. 2025 Aug;18(8):867-881. doi: 10.1016/j.jcmg.2025.04.007. Epub 2025 Jul 3. PMID 40608042
- [Background] Habibi M, Lima JA, Khurram IM, Zimmerman SL, Zipunnikov V, Fukumoto K, Spragg D, Ashikaga H, Rickard J, Marine JE, Calkins H, Nazarian S. Association of left atrial function and left atrial enhancement in patients with atrial fibrillation: cardiac magnetic resonance study. Circ Cardiovasc Imaging. 2015 Feb;8(2):e002769. doi: 10.1161/CIRCIMAGING.114.002769. PMID 25652181
- [Background] Goldberger JJ, Arora R, Green D, Greenland P, Lee DC, Lloyd-Jones DM, Markl M, Ng J, Shah SJ. Evaluating the Atrial Myopathy Underlying Atrial Fibrillation: Identifying the Arrhythmogenic and Thrombogenic Substrate. Circulation. 2015 Jul 28;132(4):278-91. doi: 10.1161/CIRCULATIONAHA.115.016795. PMID 26216085
- [Background] Kamel H, Longstreth WT Jr, Tirschwell DL, Kronmal RA, Marshall RS, Broderick JP, Aragon Garcia R, Plummer P, Sabagha N, Pauls Q, Cassarly C, Dillon CR, Di Tullio MR, Hod EA, Soliman EZ, Gladstone DJ, Healey JS, Sharma M, Chaturvedi S, Janis LS, Krishnaiah B, Nahab F, Kasner SE, Stanton RJ, Kleindorfer DO, Starr M, Winder TR, Clark WM, Miller BR, Elkind MSV; ARCADIA Investigators. Apixaban to Prevent Recurrence After Cryptogenic Stroke in Patients With Atrial Cardiopathy: The ARCADIA Randomized Clinical Trial. JAMA. 2024 Feb 20;331(7):573-581. doi: 10.1001/jama.2023.27188. PMID 38324415
- [Background] Kleindorfer DO, Towfighi A, Chaturvedi S, Cockroft KM, Gutierrez J, Lombardi-Hill D, Kamel H, Kernan WN, Kittner SJ, Leira EC, Lennon O, Meschia JF, Nguyen TN, Pollak PM, Santangeli P, Sharrief AZ, Smith SC Jr, Turan TN, Williams LS. 2021 Guideline for the Prevention of Stroke in Patients With Stroke and Transient Ischemic Attack: A Guideline From the American Heart Association/American Stroke Association. Stroke. 2021 Jul;52(7):e364-e467. doi: 10.1161/STR.0000000000000375. Epub 2021 May 24. No abstract available. PMID 34024117